CLINICAL TRIAL: NCT04723862
Title: Does Spironolactone Normalize Sleep-wake Luteinizing Hormone (LH) Pulse Frequency in Pubertal Girls With Hyperandrogenism? (CBS010)
Brief Title: Does Spironolactone Normalize Sleep-wake Luteinizing Hormone Pulse Frequency in Pubertal Girls With Hyperandrogenism?
Acronym: CBS010
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Christine Burt Solorzano, Assistant Professor in Pediatrics, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HSR200015; R01HD102060 (NIH)
Record Dates: First submitted 2020-11-18; First posted 2021-01-26 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Hyperandrogenism; Polycystic Ovary Syndrome; Puberty
Keywords: Hyperandrogenism; Polycystic ovary syndrome; Puberty
MeSH Terms: conditions — Hyperandrogenism; Polycystic Ovary Syndrome | interventions — Spironolactone

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment allocation will be double-blinded. The blind will be broken in the event of any adverse effects that would also lead to study withdrawal. The blind for a given subject will be lifted after the subject completes the study and analysis is complete for that subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spironolactone (Experimental): Prior to the first or second admission (randomly determined), participants will be pretreated for 2 weeks with spironolactone (50 mg twice daily).
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): Prior to the first or the second admission (randomly determined), participants will be pretreated for 2 weeks with placebo (twice daily).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — Spironolactone is an androgen-receptor blocker commonly used (off-label) for hyperandrogenism. The spironolactone dose will be 50 mg taken orally twice daily (for two weeks before admission to the Clinical Research Unit).
  Arms: Spironolactone
Drug: Placebo — Placebo contains only inert ingredients and is not expected to exert any direct physiological effects.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if, in mid- to late pubertal girls with hyperandrogenism (HA), androgen-receptor blockade (spironolactone) alone normalizes sleep-wake luteinizing hormone (LH) pulse frequency (primary endpoint) and overall LH and follicle-stimulating hormone secretion (secondary endpoints).

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blinded crossover study to test the following hypothesis: In mid- to late pubertal girls with hyperandrogenism, spironolactone (50 mg twice daily) for 2 weeks will reduce sleep-associated luteinizing hormone (LH) pulse frequency compared to placebo treatment. To test this hypothesis, 16 late pubertal girls (signified by either [a] post-menarcheal status [Tanner breast stages 2-5] or [b] Tanner breast stage of 4 or 5 [whether pre-menarcheal or post-menarcheal], but no more than 4 years post-menarcheal) with hyperandrogenism (serum [calculated] free testosterone concentration greater than the Tanner stage-specific reference range and/or clinical hirsutism) will undergo two clinical research unit (CRU) admissions separated by at least 4 weeks. During each admission, blood will be obtained every 10 minutes through an indwelling IV catheter from 1600 to 0700 h. This will allow full characterization of pulsatile LH secretion in addition to other hormone measurements. Formal polysomnography will be performed during CRU admissions. Subjects will be randomized to be pretreated for 2 weeks with either spironolactone (an androgen receptor blocker commonly used for hyperandrogenism) or placebo prior to the first admission; subjects will be pretreated with the other medication (placebo or spironolactone) for 2 weeks before the second admission in accordance with a cross-over design. The primary endpoint is LH pulse frequency while asleep. (LH pulse frequency while awake is an important secondary endpoint). The sleep-associated LH pulse frequency data from the spironolactone and placebo admissions will be analyzed via a hierarchical linear mixed model (HLMM). Secondary endpoints will include the relationships between sleep stages and LH pulse initiation (analyzed as per Lu et al., Neuroendocrinology 2018 [Epub ahead of print - doi: 10.1159/000488110]), and we will test the following hypothesis: In mid- to late pubertal girls with hyperandrogenism, spironolactone will enhance the ability of rapid eye movement (REM) sleep to inhibit LH pulse initiation.

ELIGIBILITY:
Inclusion Criteria:

* Mid- to late pubertal adolescent girls as signified by either (a) post-menarcheal status (Tanner breast stages 2-5) or (b) Tanner breast stage of 4 or 5 (whether pre-menarcheal or post-menarcheal) ages 10-17 years.
* Hyperandrogenism, defined as a serum (calculated) free testosterone concentration greater than the Tanner stage-specific reference range and/or clinical hirsutism
* General good health (excepting obesity, hyperandrogenism, PCOS, and adequately-treated hypothyroidism)
* Willing to strictly avoid pregnancy with use of reliable non-hormonal methods during the study period.

Exclusion Criteria:

* Inability/incapacity to provide informed consent
* Males will be excluded (hyperandrogenism is unique to females)
* Age < 10 or > 17 years (this study is designed to elucidate mechanisms underlying emerging PCOS in mid- to late pubertal adolescent girls
* Post-menarcheal by > 4 years
* Obesity resulting from a well-defined endocrinopathy, or genetic syndrome
* To ensure that blood withdrawal is within safe limits, weight < 21.5 kg is an exclusion criterion.
* Since underweight can alter pulsatile LH secretion, BMI-for-age percentile < 5 is an exclusion criterion.
* Positive pregnancy test or current lactation. Subjects with a positive pregnancy test will be informed of the result by the screening physician. Under Virginia law, parental notification is not required for minors. However, the screening physician will encourage the subject to tell her parent(s). We will counsel the adolescent about the importance of appropriate prenatal care/counseling. We will offer appropriate follow-up at the Teen Health Clinic at UVA and/or encourage the adolescent to secure prompt care via their primary care physician's office.
* Evidence for non-physiologic or non-PCOS causes of hyperandrogenism and/or anovulation
* Evidence of virilization (e.g., rapidly progressive hirsutism, deepening of the voice, clitoromegaly)
* Total testosterone > 150 ng/dl, which suggests the possibility of virilizing ovarian or adrenal tumor.
* DHEA-S elevation > 1.5 times the upper reference range limit. Mild elevations may be seen in adolescent HA and in PCOS, and will be accepted in these groups.
* Early morning 17-hydroxyprogesterone > 300 ng/dl measured in the follicular phase, which suggests the possibility of congenital adrenal hyperplasia (if elevated during the luteal phase, the 17-hydroxyprogesterone will be repeated during the follicular phase). NOTE: if a 17-hydorxyprogesterone > 300 ng/dl is confirmed on repeat testing, an ACTH stimulated 17-hydroxyprogesterone < 1000 ng/dl performed by the subject's personal physician will be required for study participation.
* Any abnormal TSH concentration will trigger repeat testing. In many cases when TSH is initially abnormal, a repeat TSH will be normal. These subjects will be permitted to continue study. If TSH remains abnormal on repeat testing, the subject will be referred to her primary medical provider. In some cases, a participant's primary medical provider will elect to simply observe a mildly low (> 0.1) or mildly elevated (< 10) if stable. In such cases, we will accept a TSH between 0.3 and 7 (inclusive) if it has remained stable for at least 6 months-such TSH values are exceedingly unlikely to influence the central reproductive axis or to influence the risks of the study. Notably, subjects with reasonably-treated primary hypothyroidism-reflected by TSH values between 0.3 and 7-on a stable dose of thyroid hormone (i.e., same dose for at least 2 months) will not be excluded.
* Prolactin concentration > 30 ng/mL (confirmed on repeat). Mild prolactin elevations may be seen in adolescents and women with HA/PCOS or obesity.
* History and/or physical exam findings suggestive of Cushing's syndrome, adrenal insufficiency, or acromegaly.
* History and/or physical exam findings suggestive of hypogonadotropic hypogonadism (e.g., symptoms of estrogen deficiency) including functional hypothalamic amenorrhea (which may be suggested by a constellation of symptoms including restrictive eating patterns, excessive exercise, psychological stress, etc.)
* Persistent hemoglobin < 11.5 g/dL for non-African American subjects; hemoglobin < 11.0 g/dL for African American subjects (confirmed on repeat). Importantly, documentation of a hemoglobin ≥ 11.0 g/dL for African American subjects or ≥ 11.5 g/dL for non-African American subjects in the month prior to the CRU admission is required for frequent sampling protocol in the CRU.
* Severe thrombocytopenia (platelets < 50,000 cells/microliter) or leukopenia (total white blood count < 4,000 cells/microliter)
* Previous diagnosis of diabetes, fasting glucose ≥ 126 mg/dl, or a hemoglobin A1c ≥ 6.5%
* Persistently abnormal sodium or potassium concentration. Bicarbonate concentrations < 20 or > 30.
* Liver test abnormalities, with two exceptions: (1) mild bilirubin elevations will be accepted in the setting of known Gilbert's syndrome or when the subject's primary care provider provides a presumptive diagnosis of Gilbert's syndrome and has no plans for further work-up; (2) mild transaminase (ALT, AST) elevations may be seen in obese/HA/PCOS girls, so stable elevations < 1.5 times the upper limit of normal will be accepted in this group.
* Absolute contraindications to spironolactone use include history of allergy to spironolactone, anuria, acute renal insufficiency, significant impairment of renal excretory function, hyperkalemia, primary adrenal insufficiency (Addison's disease), and concomitant use of eplerenone
* Significant history of cardiac or pulmonary dysfunction (e.g., known or suspected congestive heart failure, asthma requiring intermittent systemic corticosteroids, etc.)
* Decreased renal function evidenced by GFR < 60 ml/min/1.73m2
* History of cancer diagnosis and/or treatment (with the exception of basal cell or squamous cell skin carcinoma) unless they have remained clinically disease free (based on appropriate surveillance) for five years.

Ages: 10 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Sleep-Associated Luteinizing Hormone (LH) Pulse Frequency Between Admission With Spironolactone Versus Placebo | Baseline to 2 months
  The sleep-associated (22:00 h - 07:00 h) luteinizing hormone (LH) pulse frequency data from the spironolactone and placebo admissions will be analyzed via a hierarchical linear mixed model (HLMM). Sleep-associated LH pulse frequency will be compared between the spironolactone admission and the placebo admission via a linear contrast of the HLMM least squares LH pulse frequency means.

SECONDARY OUTCOMES:
Change in Wake-Associated Luteinizing Hormone (LH) Pulse Frequency Between Admission With Spironolactone Versus Placebo | Baseline to 2 months
  The wake-associated (16:00 - 22:00) luteinizing hormone (LH) pulse frequency data from the spironolactone and placebo admissions will be analyzed via a hierarchical linear mixed model (HLMM). Wake-associated LH pulse frequency will be compared between the spironolactone admission and the placebo admission via a linear contrast of the HLMM least squares LH pulse frequency means.
Change in Proportion of Luteinizing Hormone (LH) Pulses with Preceding REM Sleep With and Without Spironolactone | Baseline to 2 months
  We will analyze the proportion of luteinizing hormone (LH) pulses with REM sleep documented in the 5 minutes before each pulse and assess whether this is different between admissions with and without spironolactone. Our hypothesis is that, in the setting of hyperandrogenemia, androgen excess results in more LH pulses associated with REM sleep and that androgen blockade with spironolactone will decrease the number of LH pulses that have REM sleep immediately before the pulse. The determination of sleep stages before LH pulse initiation will be conducted as recently described by our group (Lu et al., Neuroendocrinology 2018 [Epub ahead of print - doi: 10.1159/000488110]). The differences in proportion of REM sleep-associated LH pulses between spironolactone and placebo admissions will be analyzed via a hierarchical linear mixed model (HLMM) and compared via a linear contrast of the HLMM least squares LH pulse frequency means.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Burt Solorzano, MD, Principal Investigator — University of Virginia Center for Research in Reproduction
Locations (1):
- Center for Research in Reproduction, University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No